CLINICAL TRIAL: NCT05283148
Title: Association Between Low Bone Density, Vertebral Fractures, and Pain in Sickle Cell Disease
Brief Title: Sickle Cell Disease (SCD) Bone Pain Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1782537; K23HL148310 (NIH); 2020095 (Other Grant/Funding Number: Doris Duke Charitable Foundation)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia; Low Bone Density; Osteoporosis; Osteopenia; Vertebral Fracture; Vertebral Compression; Osteonecrosis; Ischemic Necrosis; Avascular Necrosis
Keywords: sickle cell disease; sickle cell anemia; low bone density; osteoporosis; osteopenia; low bone mass
MeSH Terms: conditions — Anemia, Sickle Cell; Bone Diseases, Metabolic; Osteoporosis; Spinal Fractures; Osteonecrosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCD Bone Pain Study Cohort (Other): Prospective cohort of 50 adults with sickle cell disease (SCD) undergoing research DXA scan to assess bone mineral density and thoracolumbar morphometry for vertebral fracture analysis
  Interventions: Other: Dual-energy X-ray absorptiometry; Other: Vertebral fracture analysis; Other: Adult Sickle Cell Quality of Life Measurement System pain impact questionnaire

INTERVENTIONS:
Other: Dual-energy X-ray absorptiometry — Measure bone mineral density at the lumbar spine, left total hip, left forearm, and whole body
  Other Names: DXA scan
Other: Vertebral fracture analysis — Obtain thoracolumbar morphometry in DXA scan, then determine presence and severity of vertebral compression fractures by VFA
  Other Names: VFA
Other: Adult Sickle Cell Quality of Life Measurement System pain impact questionnaire — Calculate patient-reported total pain scores to determine the pain phenotype of each study participant
  Other Names: ASCQ-Me Pain scores

SUMMARY:
A prospective study to determine how low bone mineral density and/or vertebral compression fractures associate with pain in adults with sickle cell disease

DETAILED DESCRIPTION:
The investigators hypothesize that adults with sickle cell disease (SCD) and low bone density and/or vertebral compression fractures on a dual X-ray absorptiometry (DXA) scan (adjusted for age, sex, SCD genotype, relevant labs, presence of osteonecrosis, and SCD-modifying therapies) will report more severe pain than those with normal bone density or no vertebral fractures. The Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) is a validated patient-reported outcome measure of physical, mental, and social health in adults with SCD. This cross-sectional observational study involves obtaining a baseline DXA scan, vertebral fracture analysis (VFA) and pain assessment using ASCQ-Me pain impact scores. The investigators plan to recruit 50 adults with SCD followed at University of California Davis Medical Center between Nov 2022- Dec 2023 and anticipate enrolling up to 4 adults with SCD per month. The study endpoints are listed below:

* To determine the association between bone density Z-scores and ASCQ-Me pain impact scores in a prospective cohort of adults with SCD
* To study the association between Spine Deformity Index scores (SDI, a proxy for vertebral fracture analysis) and ASCQ-Me pain impact scores in a prospective cohort of adults with SCD
* To assess the correlation between baseline hematological and biochemical laboratory parameters (including bone biomarkers), bone density, and/or vertebral fractures in a prospective cohort of adults with SCD

The investigators' goal is to complete primary data analysis by Mar 2024. As an exploratory endpoint, 1cc of serum and 5cc of urine will be collected from each study participant once (at baseline), after an overnight fast, for bone biomarker analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years with SCD (any genotype, confirmed by hemoglobin electrophoresis or high performance liquid chromatography)
* Ability to provide written informed consent
* Ability to lay on a DXA scanner
* Negative urine pregnancy test for women of childbearing potential at study entry

Exclusion Criteria:

* Pregnant women
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Hospitalizations (any cause) within 2 weeks of study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2026-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Oyebimpe O Adesina, MD, MS, Principal Investigator — UC Davis School of Medicine
Locations (1):
- UC Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adesina O, Voutsinas JM, Wu QV, Teos LY, Rokni M, Nalbant H, Nardo L, Wun T, Zemel BS. Low bone mineral density and pain impact in adults with sickle cell disease. Blood Adv. 2025 Oct 24:bloodadvances.2025015957. doi: 10.1182/bloodadvances.2025015957. Online ahead of print. PMID 41135058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and twenty-eight unique adults (age 18 years and older) with SCD of any genotype seen in the Adult Sickle Cell clinic at UCD's Comprehensive Cancer Center between 2022-2023 were eligible to participate in the SCD Bone Pain study.
Pre-assignment Details: From this convenience sample of 128 SCD adults, 72 were approached to participate in the study, and 53 participants eventually enrolled in the SCD Bone Pain study
Groups:
- SCD Bone Pain Study Cohort: The SCD Bone Pain study was a single-arm, prospective, observational cohort study of 53 adults with sickle cell disease (SCD) undergoing research DXA scans to assess bone mineral density, thoracolumbar morphometry for vertebral fracture analyses, and ASC-Me pain impact assessment.
  Definitions:
  Dual-energy X-ray absorptiometry (DXA) scan: Used to measure bone mineral density at the lumbar spine, total hip, forearm, and whole body
  Vertebral fracture analysis (VFA): Obtained from thoracolumbar morphometry in DXA scanner, then grade presence and severity of vertebral compression fractures using spinal deformity index
  Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) pain impact questionnaire: Calculate patient-reported total pain scores to determine the pain phenotype of each study participant
Period: Overall Study
Arm/Group | SCD Bone Pain Study Cohort
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- SCD Bone Pain Study Cohort: Prospective cohort of 53 adults with sickle cell disease (SCD) to assess the following:
  1. Bone mineral density (BMD) at the lumbar spine, left total hip, left forearm, and whole body, using a dual-energy X-ray absorptiometry (DXA) scan
  2. Spinal deformity index (measure of presence and severity of vertebral fractures) using thoracolumbar morphometry obtained from the DXA scanner
  3. Patient-reported pain impact score obtained from the Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) Pain impact questionnaire
Arm/Group | SCD Bone Pain Study Cohort
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: Years] — Age (years) at study visit date
  Years | 36 [20 to 67]
Sex: Female, Male [Count of Participants; unit: Participants] — Patient-reported sex (at birth) obtained on study visit date
  Participants
    Female | 34
    Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 50
  White | 1
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 53
Height [Median (Full Range); unit: cm] — Participant height measured on study visit date
  cm | 172 [152 to 194]
Body mass index (BMI) [Median (Full Range); unit: kg/m2] — BMI as of study visit date
  kg/m2 | 24.6 [18.7 to 39.9]
Sickle cell disease (SCD) genotype [Count of Participants; unit: Participants] — SCD genotype confirmed by hemoglobin electrophoresis or hemoglobin analysis
  Participants
    Hb SS | 30
    Hb SC | 15
    Hb SB0 | 5
    Hb SB+ | 2
    Hb SD | 1
Osteonecrosis [Count of Participants; unit: Participants] — Number of participants with radiographically confirmed osteonecrosis at study entry
  Participants
    Yes | 22
    No | 31

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density
Description: Areal bone mineral density of the lumbar spine measured by dual-energy X-ray absorptiometry (DXA) scan and reported in grams per square centimeter.
Time Frame: Baseline
Measure: Median (Full Range); unit: g/cm2
Groups:
- Group A: Female participants
- Group B: Male Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 34 | 19
g/cm2 | 0.97 [0.62 to 1.31] | 1.0 [0.72 to 1.67]
Statistical Analysis 1: Comparison: Group A vs Group B; Comparison between Group A and Group B as defined above. Values are reported as median (full range) for each group, measured by DXA at the lumbar spine. Distribution was non-normal, so a Wilcoxon rank-sum test (two-sided) was used. A p-value < 0.05 was considered statistically significant; Test type: Other — Distribution was non-normal, so a Wilcoxon rank-sum test (two-sided) was used; p = 0.321, Wilcoxon rank-sum test (two-sided) — A p-value < 0.05 was considered statistically significant

2. Primary Outcome: Lumbar Spine Bone Mineral Density-Z-scores
Description: Number of standard deviations between measured lumbar spine bone mineral density (g/cm2) for each participant and mean lumbar spine bone mineral density (g/cm2) of the reference population. A Z-score of 0 represents the mean of the reference population. A negative Z-score means the measured bone mineral density values are lower (worse) the reference mean, while positive Z-scores mean they are above/higher. Bone mineral density Z-scores ≤ -2 indicates low bone density.
Time Frame: Baseline
Measure: Median (Full Range); unit: Z-score
Arm/Group | Group A | Group B
Number analyzed (Participants) | 34 | 19
Z-score | -1.35 [-4.40 to 1.60] | -1.60 [-4.30 to 4.30]
Statistical Analysis 1: Comparison: Group A vs Group B; Comparison between Group A and Group B as defined above. Values are reported as median ± full range for each group, derived from DXA lumbar spine scans. Welch two-sample t-test (two-sided) was used to account for unequal variances. A p-value < 0.05 was considered statistically significant; Test type: Other — Welch two-sample t-test (two-sided) was used to account for unequal variances; p = 0.714, Welch two sample t-test — A p-value < 0.05 was considered statistically significant

3. Primary Outcome: Total Hip Bone Mineral Density (BMD)
Description: Areal bone mineral density of the total hip measured by dual-energy X-ray absorptiometry (DXA) scan and reported in grams per square centimeter.
Time Frame: Baseline
Measure: Median (Full Range); unit: g/cm2
Arm/Group | Group A | Group B
Number analyzed (Participants) | 34 | 19
g/cm2 | 0.90 [0.66 to 1.34] | 1.03 [0.67 to 1.76]
Statistical Analysis 1: Comparison: Group A vs Group B; Comparison between Group A and Group B as defined above. Values are reported as median (full range) for each group, measured by DXA at the total hip. Distribution was non-normal, so a Wilcoxon rank-sum test (two-sided) was used. A p-value < 0.05 was considered statistically significant; Test type: Other — Distribution was non-normal, so a Wilcoxon rank-sum test (two-sided) was used; p = 0.09, Wilcoxon rank-sum test (two-sided) — p-value < 0.05 was considered statistically significant

4. Primary Outcome: Total Hip Bone Mineral Density-Z-scores
Description: Number of standard deviations between measured total hip bone mineral density (g/cm2) for each participant and mean total hip bone mineral density (g/cm2) of the reference population. A Z-score of 0 represents the mean of the reference population. A negative Z-score means the measured bone mineral density values are lower (worse) the reference mean, while positive Z-scores mean they are above/higher. Bone mineral density Z-scores ≤ -2 indicates low bone density.
Time Frame: At enrollment
Measure: Median (Full Range); unit: Z-score
Arm/Group | Group A | Group B
Number analyzed (Participants) | 34 | 19
Z-score | -0.75 [-2.30 to 2.00] | -0.5 [-2.7 to 3.5]
Statistical Analysis 1: Comparison: Group A vs Group B; Comparison between Group A and Group B as defined above. Values are reported as median ± full range for each group, derived from DXA total hip scans. Welch two-sample t-test (two-sided) was used to account for unequal variances. A p-value < 0.05 was considered statistically significant; Test type: Other — Welch two-sample t-test (two-sided) was used to account for unequal variances; p = 0.604, Welch two sample t-test (two sided) — A p-value < 0.05 was considered statistically significant

5. Primary Outcome: Femoral Neck Bone Mineral Density (BMD)
Description: Areal bone mineral density of the femoral neck measured by dual-energy X-ray absorptiometry (DXA) scan and reported in grams per square centimeter.
Time Frame: Baseline
Measure: Median (Full Range); unit: g/cm2
Arm/Group | Group A | Group B
Number analyzed (Participants) | 34 | 19
g/cm2 | 0.77 [0.53 to 1.30] | 0.94 [0.63 to 1.68]
Statistical Analysis 1: Comparison: Group A vs Group B; Comparison between Group A and Group B as defined above. Values are reported as median (full range) for each group, measured by DXA at the femoral neck. Distribution was non-normal, so a Wilcoxon rank-sum test (two-sided) was used. A p-value < 0.05 was considered statistically significant; Test type: Other — Distribution was non-normal, so a Wilcoxon rank-sum test (two-sided) was used; p = 0.013, Wilcoxon rank-sum test (two-sided) — A p-value < 0.05 was considered statistically significant

6. Primary Outcome: Femoral Neck Bone Mineral Density Z-scores
Description: as for outcome 2
Time Frame: Baseline
Measure: Median (Full Range); unit: Z-score
Arm/Group | Group A | Group B
Number analyzed (Participants) | 34 | 19
Z-score | -0.95 [-2.7 to 2.4] | -0.60 [-2.3 to 4.0]
Statistical Analysis 1: Comparison: Group A vs Group B; Comparison between Group A and Group B as defined above. Values are reported as median ± full range for each group, derived from DXA femoral neck scans. Welch two-sample t-test (two-sided) was used to account for unequal variances. A p-value < 0.05 was considered statistically significant; Test type: Other — Welch two-sample t-test (two-sided) was used to account for unequal variances; p = 0.166, Welch two sample t-test — A p-value < 0.05 was considered statistically significant

7. Primary Outcome: Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) Pain Impact T-scores
Description: Patient-reported outcome measure of pain impact in the preceding 7 days before bone density measurements. The Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) pain impact T-scores range from about 30-100. The ASCQ-Me pain impact T-score has standardized mean T-score of 50 and standard deviation of 10, which were derived from a reference population of ambulatory adult with sickle cell disease across the United States. ASCQ-Me pain impact T-scores less than 50 are lower/worse than the reference mean (more severe pain impact), while pain impact T-scores greater than 50 are above/better than the reference mean (less severe pain impact)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: T-score
Groups:
- Group A: Low bone mineral density (Z-score ≤ -2.0) at baseline
- Group B: Normal bone mineral density (Z-score > -2.0) at baseline
Arm/Group | Group A | Group B
Number analyzed (Participants) | 23 | 30
T-score | 47.1 [42.4 to 52.8] | 52.4 [45.3 to 56.5]
Statistical Analysis 1: Comparison: Group A vs Group B; Comparison between Group A and Group B as defined above. Values are reported as median (interquartile range) for each group, based on the ASCQ-Me Pain Impact instrument (lower scores indicate worse pain impact). Welch two-sample t-test (two-sided) was used to account for unequal variances. A p-value < 0.05 was considered statistically significant; Test type: Other — Welch two-sample t-test (two-sided) was used to account for unequal variances; p = 0.23, Welch two sample t-test (two sided) — A p-value < 0.05 was considered statistically significant

8. Secondary Outcome: Spinal Deformity Index
Description: The spinal deformity index (SDI) is a semi-quantitative measure of number and severity of vertebral fractures observed on lateral spine X-rays of the thoracolumbar spine. To calculate the SDI, vertebrae are assigned a score as follows: 0 (no fracture), 1 (mild fracture), 2 (moderate fracture), and 3 (severe fracture). The total SDI is the summation of all T12-L4 vertebrae measured on the lateral spine X-rays. Minimum SDI =0 and Maximum SDI=15. Higher scores mean increased (worse) fracture burden, lower scores mean decreased (less) fracture burden.
Time Frame: Baseline
Population: Statistical analysis of spinal deformity index is ongoing. Complete results will be provided by February 2026.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 23 | 30
score on a scale | 2.00 (2.71) | 3.13 (3.98)

ADVERSE EVENTS:
Time Frame: 13 months
Groups:
- SCD Bone Pain Study Cohort: Prospective cohort of 53 adults with sickle cell disease (SCD) undergoing research DXA scan to assess bone mineral density and thoracolumbar morphometry for vertebral fracture analysis
  Dual-energy X-ray absorptiometry: Measure bone mineral density at the lumbar spine, left total hip, left forearm, and whole body
  Vertebral fracture analysis: Obtain thoracolumbar morphometry in DXA scan, then determine presence and severity of vertebral compression fractures by VFA
  Adult Sickle Cell Quality of Life Measurement System pain impact questionnaire: Calculate patient-reported total pain scores to determine the pain phenotype of each study participant
Arm/Group | SCD Bone Pain Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

LIMITATIONS AND CAVEATS:
This prospective study on the association between bone density and pain in SCD is limited by its cross-sectional study design and small sample size. We can only report associations between the predictor variables and outcomes of interest, not causality. Since joint imaging was only done based on symptoms, we may have missed participants with asymptomatic osteonecrosis. Lastly, DXA scans are widely used to clinically assess severe low BMD but cannot differentiate trabecular vs cortical bone loss.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT05283148/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT05283148/ICF_001.pdf